CLINICAL TRIAL: NCT03108131
Title: A Phase II, Open-Label, Single-Arm, Multi-Cohort, Proof-of-Principle Study to Investigate the Efficacy of Cobimetinib and Atezolizumab in Advanced Rare Tumors
Brief Title: Cobimetinib and Atezolizumab in Treating Participants With Advanced or Refractory Rare Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0869; NCI-2018-01399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0869 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Skin Squamous Cell Carcinoma; Appendix Adenocarcinoma; Rare Lesion; Locally Advanced Malignant Neoplasm; Locally Advanced Skin Squamous Cell Carcinoma; Metastatic Malignant Neoplasm; Metastatic Skin Squamous Cell Carcinoma; Metastatic Small Intestinal Adenocarcinoma; Rare Neoplastic Syndrome; Refractory Malignant Neoplasm; Stage IV Small Intestinal Adenocarcinoma AJCC v8; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Adenocarcinoma, Mucinous; Neoplasm Metastasis; Neoplasms | interventions — atezolizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cobimetinib, atezolizumab) (Experimental): Participants receive cobimetinib PO QD on days 1-21 and atezolizumab IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518

SUMMARY:
This phase II trial studies how well cobimetinib and atezolizumab work in treating participants with rare tumors that have spread to other places in the body (advanced) or that does not respond to treatment (refractory). Cobimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cobimetinib and atezolizumab may work better in treating participants with advanced or refractory rare tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of cobimetinib plus atezolizumab (COTEZO) in cohorts of advanced rare tumors using objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS) on COTEZO in cohorts of advanced rare tumors per RECIST v1.1 and immune-related (ir)RECIST.

II. To determine overall survival (OS) on COTEZO in cohorts of advanced rare tumors.

III. To determine disease control rate (DCR) and duration of response (DOR) on COTEZO in cohorts of advanced rare tumors per RECIST v1.1 and irRECIST.

IV. To determine objective response rate (ORR) per immune-related RECIST criteria.

V. To determine safety profile and adverse events encountered by patients with advanced rare tumors treated with COTEZO.

VI. To collect and bank tumor tissue and peripheral blood for future correlative analyses from patients with advanced rare tumors treated with COTEZO.

OUTLINE:

Participants receive cobimetinib orally (PO) once daily (QD) on days 1-21 and atezolizumab intravenously (IV) over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants followed up every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and must be willing to give written informed consent in accordance with institutional and federal guidelines. Patients must be able to comply with the requirements and assessments of the study protocol
* Must have histologically or cytologically documented rare tumor as defined per protocol that is metastatic or locally advanced and unresectable. Patients with locally advanced cutaneous squamous cell carcinoma that are technically resectable but in whom surgery is expected to lead to substantial function impairment or disfigurement are eligible
* Must be refractory or intolerant to standard lines of therapy
* Must have completed prior chemotherapy, immunotherapy, or radiation therapy at least 14 days prior to start of treatment and all toxicity must be resolved to Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grade 1 (with the exception of CTCAE v4.0 grade 2 neuropathy) prior to start of treatment
* Presence of radiographically evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Tissue Parameters: a. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks are preferred) or at least 4 unstained slides, with an associated pathology report, for testing of tumor PD-L1 expression (tumor tissue from bone metastases is not evaluable for PD-L1 expression and is therefore not acceptable). b. Tumor tissue should be of good quality based on total and viable tumor content. Fine needle aspiration, brushing, cell pellet from pleural effusion, bone metastases, and lavage samples are not acceptable. For core-needle biopsy specimens, at least three cores should be submitted for evaluation. c. Patients who do not have tissue specimens meeting eligibility requirements must be willing to undergo a biopsy during the screening period
* Absolute neutrophil count (ANC) >= 1,000/mcL (obtained within 14 days prior to enrollment)
* Platelets >= 75,000/mcL (obtained within 14 days prior to enrollment)
* Hemoglobin >= 9 g/dL (obtained within 14 days prior to enrollment)
* Calculated creatinine clearance > 30 ml/min (obtained within 14 days prior to enrollment)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 3 x institutional upper limit of normal (IULN) without liver mets or =< 5 x IULN with liver metastases (obtained within 14 days prior to enrollment)
* Bilirubin =< 1.5 mg/dL (obtained within 14 days prior to enrollment)
* Able to swallow pills
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for >= 1 year
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (e.g., implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception)
* For individual baskets:

  * Appendiceal adenocarcinoma

    * Not considered candidate for curative surgery
  * Cutaneous squamous cell carcinoma

    * Patients with either metastatic or locally advanced cutaneous squamous cell carcinoma that are technically resectable but in whom surgery is expected to lead to substantial function impairment or disfigurement are eligible
  * Small bowel adenocarcinoma

    * Must be refractory or intolerant to at least one line of fluorouracil (5FU)-based chemotherapy for metastatic disease

Exclusion Criteria:

* Presence of brain metastases (unless they have been adequately treated with radiotherapy or surgery and stable for at least 30 days prior to enrollment provided patient is neurologically asymptomatic and without corticosteroid treatment for at least 7 days prior to enrollment)
* Uncontrolled intercurrent illness including, but not limited to diabetes, hypertension, severe infection, severe malnutrition, unstable angina, class III-IV New York Heart Association (NYHA) congestive heart failure, ventricular arrhythmias, active ischemic heart disease, or myocardial infarction within 6 months prior to enrollment
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration
* Patients will be excluded from study participation if they currently are known to have any of the following risk factors for RVO: a. Glaucoma with intraocular pressure >= 21 mmHg b. Grade >= 2 serum cholesterol c. Grade >= 2 hypertriglyceridemia d. Grade >= 2 or symptomatic hyperglycemia (fasting) e. Grade >= 2 uncontrolled hypertension (patients with a history of hypertension controlled with anti-hypertensive medication to grade =< 1 are eligible)
* Active malignancy (other than colorectal carcinoma [CRC]) or a history of prior malignancy within the past 3 years. Adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, ductal carcinoma in situ, other low grade lesions such as incidental appendix carcinoid, or any other cancer from which the patient has been disease and treatment free for two years are allowed. Prostate cancer patients on active surveillance are eligible
* Pregnant or nursing patients due to risk of fetal or nursing infant harm. Women/men of reproductive potential who do not agree to use an effective contraceptive method while on study and for at least 6 months after study treatment
* Exclusion criteria related to study medication (any cancer immunotherapy including CD137 agonists, anti-PD-1, anti-PD-L1, or anti-CTLA4 or any MEK or ERK inhibitor)
* Left ventricular ejection fraction (LVEF) < institutional lower limit of normal or < 50%
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis a. Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. b. Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible. c. Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* History of human immunodeficiency virus (HIV) infection or active hepatitis B (chronic or acute) or hepatitis C infection. a. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. b. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Active tuberculosis or severe infections within 4 weeks prior to cycle 1, day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with systemic immuno-stimulatory agents (including but not limited to interferon [IFN] or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to cycle 1, day 1
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* For individual baskets:

  * Appendiceal adenocarcinoma

    * Must not have clinically symptomatic malignant bowel obstruction
  * Cutaneous squamous cell carcinoma

    * None
  * Small bowel adenocarcinoma

    * Must not have clinically symptomatic malignant small bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal P Raghav, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 49 patients that was enrolled at MD Anderson Cancer Center Houston, Tx, only 20 patients had Small Bowel Adenocarcinoma. The rest had other solid tumors and their data was not used in the analysis for the group of patients with Small Bowel Adenocarcinoma.
Groups:
- Small Bowel Adenocarcinoma: Must be refractory or intolerant to at least one line of 5FU-based chemotherapy for metastatic disease and must not have clinically symptomatic malignant small bowel obstruction. Cobimetinib (60 mgorally once daily for days 1 - 21) and atezolizumab (840 mg intravenously every 2 weeks) every 28-day cycle.
Period: Overall Study
Arm/Group | Small Bowel Adenocarcinoma
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: To evaluate the efficacy of cobimetinib plus atezolizumab (COTEZO) in cohorts of advanced rare tumors using objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Efficacy as determined by complete response and partial response.
Time Frame: Patient will be on study up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 20
Participants | 2

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) includes patients with tumor maintained at Stable Disease (SD), Partial Response (PR) and Complete Response (CR).
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 20
percentage of participants | 45 [23.1 to 68.5]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from randomization until first evidence of disease progression or death
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 20
months | 2.4 [1.3 to 3.5]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to death
Time Frame: 3 years
Population: 2 of the patients was not included in the analysis of PFS because their surgical cancellations were unrelated to progressive disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 18
months | 8.8 [5.6 to 12]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Small Bowel Adenocarcinoma
All-Cause Mortality (participants affected / at risk) | 9/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Small Bowel Adenocarcinoma (N=20)
Anemia (Blood and lymphatic system disorders) | 8
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Retinopathy (Eye disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Dry Mouth (Gastrointestinal disorders) | 1
Gatroesophageal Disease (Gastrointestinal disorders) | 1
Gastrointestinal Disease-Others (Sore Gums) (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Limb Edema (General disorders) | 3
Fatigue (General disorders) | 9
Fever (General disorders) | 2
Gait Disturbances (General disorders) | 1
UTI (Infections and infestations) | 3
Infections and Infestations-Other (Influenza A and H1 2009 (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Alanin aminotransferace increase (Investigations) | 4
Alkaline Phosphatase increase (Investigations) | 5
Aspartate aminotransferase Increase (Investigations) | 5
Total Bilirubin Increase (Investigations) | 1
Cholesterol High (Investigations) | 2
CPK Increased (Investigations) | 6
INR increased (Investigations) | 1
Platelet Count decrease (Investigations) | 1
White Blood Cell Count Increaese (Investigations) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Nervous System Disorders-others (Brain Metastasis) (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-planter Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03108131/Prot_SAP_000.pdf